CLINICAL TRIAL: NCT05294211
Title: Marani Prenatal Connected Care (M•Care) Safety and Effectiveness Study
Brief Title: Safety and Performance of a Fetal Monitoring System
Acronym: M•CARE SE
Status: Completed | Type: Interventional
Sponsor: Marani Health (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MH-001
Record Dates: First submitted 2022-03-15; First posted 2022-03-24 (Actual); Results first posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-01

CONDITIONS: Pregnancy
Keywords: antenatal monitoring; fetal monitoring
MeSH Terms: interventions — Cardiotocography

STUDY DESIGN:
Oversight: Unapproved Device: Yes

ARMS (1):
- M•care™ System + CTG (Experimental): The M•care System and standard of care CTG (cardiotocography) will be applied for fetal and maternal monitoring
  Interventions: Device: M•care™ System; Device: Cardiotocography (CTG)

INTERVENTIONS:
Device: M•care™ System — The M•care™ System will be applied for monitoring of fetal heart rate (FHR), maternal heart rate (MHR) and uterine activity (UA)
Device: Cardiotocography (CTG) — A standard of care CTG device will be applied for monitoring of fetal heart rate (FHR), maternal heart rate (MHR) and uterine activity (UA)

SUMMARY:
The objective of this study is to demonstrate the safety and performance of the M•care™ System for use in antenatal monitoring of pregnant women ≥ 32 weeks' gestation.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent and follow study instructions
* 18 years of age or older
* Pregnant subjects ≥ 32 weeks' gestation
* Singleton pregnancy
* BMI ≥15, pre-pregnancy
* BMI ≤45, pre-pregnancy
* Belly circumference ≥80 cm and ≤ 130 cm

Exclusion Criteria:

* Known major fetal malformation or chromosome abnormality
* Abdominal medical skin conditions, including surgical incisions, open wounds with our without infections, edema, or irritation
* Participants with implanted electronic devices (pacemakers, defibrillator, etc.)
* Involvement in another clinical trial currently or previously in this pregnancy that, in the investigator's opinion, would affect the conduct of this study
* Medical or obstetric problem that in the investigator's opinion would make the participant incapable of taking part in the study
* In the investigator's opinion, the participant is not likely to be available for the minimum 60 minutes of the monitoring session
* History of skin allergies to cosmetics and lotions
* Known allergies to silver, nylon, or polyester

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-01-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- NorthShore University Health System, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- M•Care™ System + CTG: Single-arm study: All subjects were monitored with both the M•wrap and the CTG reference device simultaneously for fetal heart rate (FHR), maternal heart rate (MHR), and uterine contractions (UC)
  After enrollment, the presence of FHR and MHR was confirmed by completing a 5-minute monitoring session with the M•care System.
  If a valid signal was detected, a 30-minute session was initiated in which both systems (M•care and CTG) simultaneously recorded FHR, MHR, and UC data. Up to four monitoring sessions were completed depending on the availability of the subject.
Period: Overall Study
Arm/Group | M•Care™ System + CTG
Started | 120
Completed | 80
Not Completed | 40
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 2
Not completed — Progressed to active labor | 1
Not completed — Did not complete 5-minute monitoring session | 15
Not completed — Did not have ≥ 1 minute of concurrent data | 19

BASELINE CHARACTERISTICS:
Population: Performance evaluable population, as defined by the population of subjects who had at least one minute of concurrent data collection with both devices (M•care and CTG) and did not have any major protocol violations.
Arm/Group | M•Care™ System + CTG
Number analyzed (Participants) | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 80
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 72
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 62
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 80

OUTCOME MEASURES:

1. Primary Outcome: Fetal Heart Rate (FHR)
Description: FHR as measured by the M•care System versus standard of care CTG device
Time Frame: Up to 120 minutes
Population: The performance evaluable population was defined as the population of subjects who had at least one minute of concurrent data collection with both devices (M•care and CTG) and did not have any major protocol violations. Of the 80 subjects in the performance evaluable population, no FHR data are available for one subject.
Measure: Mean (Standard Deviation); unit: BPM
Groups:
- M•Care™ System: The M•care System was applied for fetal and maternal monitoring
- Cardiotocography (CTG): A Philips Avalon FM30 or FM50 (CTG) was applied for fetal and maternal monitoring
Arm/Group | M•Care™ System | Cardiotocography (CTG)
Number analyzed (Participants) | 79 | 79
BPM | 140.1 (11.4) | 140.0 (10.7)

2. Primary Outcome: Maternal Heart Rate (MHR)
Description: MHR as measured by the M•care System versus standard of care CTG device
Time Frame: Up to 120 minutes
Population: The performance evaluable population was defined as the population of subjects who had at least one minute of concurrent data collection with both devices (M•care and CTG) and did not have any major protocol violations. Of the 80 subjects in the performance evaluable population, no MHR data are available for one subject.
Measure: Mean (Standard Deviation); unit: BPM
Arm/Group | M•Care™ System | Cardiotocography (CTG)
Number analyzed (Participants) | 79 | 79
BPM | 83.4 (12.0) | 83.1 (12.1)

3. Secondary Outcome: Uterine Contractions (UC)
Description: UC sensitivity as measured by the M•care System versus standard of care CTG device, where sensitivity is defined as the proportion of UC events identified by standard of care that are simultaneously identified by the M•care System (positive agreement).
Time Frame: Up to 120 minutes
Population: Of the 80 subjects in the performance evaluable population, no uterine contraction (UC) data are available for two subjects.
  To compare sensitivity (positive agreement) in UC events between M•care and standard of care, bootstrap resampling techniques were used to account for the correlation among repeated UC measurements within subjects. Results for the M•care System and CTG are combined due to the outcome measure of UC sensitivity (positive agreement).
Measure: Number (95% Confidence Interval); unit: proportion of true positives
Groups:
- M•Care™ System + CTG: The M•care System and standard of care CTG (cardiotocography) will be applied for monitoring uterine activity
Arm/Group | M•Care™ System + CTG
Number analyzed (Participants) | 78
proportion of true positives | 0.57 [0.50 to 0.63]

ADVERSE EVENTS:
Time Frame: 3 hours
Description: ISO 14155:2020 definitions of adverse event and serious adverse event were used.
Arm/Group | M•Care™ System + CTG
All-Cause Mortality (participants affected / at risk) | 0/120
Serious Adverse Events (participants affected / at risk) | 0/120
Other Adverse Events (participants affected / at risk) | 1/120
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | M•Care™ System + CTG (N=120)
erythema (Skin and subcutaneous tissue disorders) | 1 (1) — Mild erythema and skin irritation occurred after applying the exfoliating agent, prior to the use of the M•care System

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT05294211/Prot_SAP_000.pdf